CLINICAL TRIAL: NCT00003674
Title: Phase III Double-Blind Trial Comparing Low-Molecular Weight Heparin (LMWH) Versus Placebo in Patients With Advanced Cancer
Brief Title: Standard Therapy With or Without Dalteparin in Treating Patients With Advanced Breast, Lung, Colorectal, or Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCCTG-979251; CDR0000066775 (Registry Identifier: PDQ (Physician Data Query)); NCI-P98-0139
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer; Prostate Cancer; Veno-occlusive Disease
Keywords: stage IV colon cancer; stage IV breast cancer; recurrent breast cancer; recurrent non-small cell lung cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; stage IV prostate cancer; recurrent prostate cancer; stage IV non-small cell lung cancer; veno-occlusive disease
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Rectal Neoplasms; Small Cell Lung Carcinoma | interventions — Dalteparin; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dalteparin + standard therapy (Experimental): Patients receive dalteparin by subcutaneous injection once daily plus standard therapy. Treatment continues for 1 year in the absence of disease progression and unacceptable toxicity. Quality of life is assessed before treatment, then every month for the first year, and then every 3 months for 2 years. Patients are followed monthly for 1 year, then every 3 months for 2 years.
  Interventions: Drug: dalteparin; Drug: standard therapy
- standard therapy (Active Comparator): Patients receive standard therapy alone. Treatment continues for 1 year in the absence of disease progression and unacceptable toxicity. Quality of life is assessed before treatment, then every month for the first year, and then every 3 months for 2 years. Patients are followed monthly for 1 year, then every 3 months for 2 years.
  Interventions: Drug: standard therapy

INTERVENTIONS:
Drug: dalteparin
  Arms: dalteparin + standard therapy
Drug: standard therapy

SUMMARY:
RATIONALE: Dalteparin may be effective in inhibiting the growth of blood vessels in tumors, decreasing the risk of metastatic cancer, preventing the formation of blood clots, and improving quality of life in treating patients with advanced cancer that has not responded to previous treatment. It is not yet known if standard therapy is more effective with or without dalteparin in treating advanced breast, lung, colorectal, and prostate cancer.

PURPOSE: Randomized double blinded phase III trial to compare the effectiveness of standard therapy with or without dalteparin in treating patients who have advanced breast, lung, colorectal, or prostate cancer that has not responded to previous chemotherapy or hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effect of low molecular weight heparin (dalteparin) plus standard therapy versus standard therapy alone on the overall survival rate of patients with advanced cancers. II. Compare the toxic effects of these regimens and the effect on the quality of life of these patients. III. Assess the incidence of symptomatic thrombotic events such as deep venous thrombosis (DVT), pulmonary embolus (PE), and clotted catheters in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to prognostic index (good vs bad vs unsure), current therapy (systemic vs radiation vs both vs none), age (50 or under vs over 50), disease site (breast vs colon vs small cell lung vs nonsmall cell lung vs prostate), history of prior thrombotic event over 1 year ago (yes vs no), and gender. Patients are randomized to receive low molecular weight heparin (dalteparin) plus standard therapy or standard therapy alone.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven breast, lung, colorectal, or prostate cancer that has failed prior chemotherapy or hormone therapy No active CNS metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3500/mm3 Platelet count at least 150,000/mm3 Fibrinogen above lower limits of normal Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 3 times ULN Prothrombin time no greater than 1.5 times ULN Active partial thromboplastin time no greater than 1.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Other: No history of heparin associated thrombocytopenia At least 1 year since prior thromboembolic phenomenon such as deep venous thrombosis, pulmonary embolus, or clotted catheter No prior intolerance of unfractionated or low molecular weight heparin

PRIOR CONCURRENT THERAPY: No concurrent anticoagulation therapy No concurrent enrollment on systemic or radiation therapy study (therapy off study allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 1998-12; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | Up to 5 years

SECONDARY OUTCOMES:
Overall quality of life | Up to 5 years
Assess the incidence of symptomatic thrombotic events such as deep venous thrombosis (DVT), pulmonary embolus (PE), and clotted catheters | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Okuno, MD, Study Chair — Mayo Clinic
Locations (20):
- United States (19):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada